CLINICAL TRIAL: NCT01178060
Title: The Effectiveness of Personalized Stroke Risk Communication - A Pilot Randomized Controlled Trial
Brief Title: The Effectiveness of Personalized Stroke Risk Communication
Acronym: RiskCom
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Durham VA Medical Center (U.S. Federal Agency)
Responsible Party: Hayden Bosworth, PhD/Associate Director HSR&D and Benjamin Powers, MD/Co-I, Durham VA Medical Center
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Health Services Research
Other Study IDs: RRP 08-240
Record Dates: First submitted 2010-08-06; First posted 2010-08-09 (Estimated); Last update posted 2010-08-23 (Estimated); Status verified 2010-08

CONDITIONS: Cardiovascular Disease; Stroke
Keywords: Stroke; Risk; Communication; Cardiovascular Disease Knowledge; Improve Risk Communication
MeSH Terms: conditions — Cardiovascular Diseases; Stroke; Communication

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Personalized Risk Information (Active Comparator): Patients received personalized stroke and heart attack risk assessment information.
  Interventions: Other: Personalized Heart Attack and Stroke Risk
- Standard Education (Other): Patients received general risk information on heart attack and stroke.
  Interventions: Other: Standard Education

INTERVENTIONS:
Other: Personalized Heart Attack and Stroke Risk — Personalized assessment of heart attack and stroke risk based on 10yr predictors with individual risk factors.
  Arms: Personalized Risk Information
Other: Standard Education — Patients received a general handout describing risk factors for heart attack and stroke.
  Arms: Standard Education

SUMMARY:
The goal of this research is to improve communication to Veterans. The investigators want to improve how doctors and nurses talk to patients about the risk of heart attack and stroke. The investigators will give everyone in the study information about the risk for heart attack or stroke. The investigators will also provide information on how to reduce this risk. This information will be given in one of two ways. The investigators want to see which way of giving information works better for veterans. The investigators also want to assess the impact of personalized stroke risk communication to patients at risk for stroke on patient knowledge, beliefs, and preferences for risk reduction behaviors and evaluate the impact of personalized risk communication on medication adherence and blood pressure. The investigators plan to enroll approximately 100 veterans for this study. All veterans will be from the Durham VA Primary Care Clinics. The investigators will ask everyone to be in the study for 3 months.

DETAILED DESCRIPTION:
Background:

In 2005, over 17,000 patients were treated for stroke within the VA with a cost of almost $315 million. Prevention of stroke through reduction of established risk factors is an essential part of the VA Stroke QUERI strategic plan for the VA. In spite of this, in the Veterans Affairs, only 13% of patients with known CVD achieve target BP and cholesterol control. Combining risk factors into a composite measure of risk offers a better global assessment of individual risk and is recommended by the American Heart Association and American Stroke Association for prioritizing interventions. This practice is rarely done in routine clinical practice and its use as a tool to motivate patient behavior has not been tested. Current evidence from VA patients suggests that patients with hypertension do not adequately translate their risk factors into an accurate estimation of stroke risk. Improving the accuracy of stroke risk perceptions may be particularly important in motivating risk reduction in patients.

Objectives:

The objectives of this study are to: 1.) Assess the impact of personalized stroke risk communication to patients at risk for stroke on patient knowledge, beliefs, and preferences for risk reduction behaviors. 2.) Evaluate the impact of personalized risk communication on medication adherence and blood pressure. 3.) Explore the feasibility and obtain sample size estimates for a larger, investigator initiative research (IIR) application testing this tool.

Methods:

A two-group randomized controlled trial testing a personalized risk communication intervention compared to an education-only control group was conducted. Eighty-nine patients were randomized and followed for 3months. Both groups received written and verbal patient education on stroke risk factors and prevention. Patients in the intervention arm also received personalized risk communication based on the Framingham stroke and coronary heart disease risk scores. A verbal and graphic presentation of their personal risk, risk relative to an age matched cohort, and their optimal or target risk based on optimal risk factor modification was presented. Outcomes measured immediately following the intervention and at 3months included: risk perception and worry; risk factor knowledge; decision preference and conflict; medication adherence; health behaviors; and blood pressure.

Status:

The study finished enrollment and all follow-up visits have been completed. The data from this project is being analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Enrolled in a Durham VA Primary Care Clinic for at least one year
* Age ≥ 55 years old
* Diagnosis ICD 401.0, 401.1, or 401.9 on outpatient electronic encounter forms in the prior year
* Received a prescription for hypertensive medication (ACE inhibitors, beta blockers, calcium channel blockers, diuretics, alpha1 blockers, and/or central alpha2 agonists) in the previous year
* Inadequate BP control based on an average of prior 12-month clinic BP measurements
* Have a baseline EKG within the last 5 years to evaluate the presence of left ventricular hypertrophy.

Exclusion Criteria:

* Hospitalized at the DVAMC for a myocardial infarction (MI), coronary artery revascularization, or diagnosis of metastatic cancer in the past 6 months
* Prior history of stroke
* Active diagnosis of psychosis or dementia documented in medical record
* Participating in another chronic disease self-management study
* Resident of a nursing home
* Does not have access to a telephone
* Refusal to provide informed consent

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2008-09; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Impact of personalized risk information | baseline
  Assess the impact of personalized risk communication to patients at risk for stroke on patient knowledge, beliefs, and preferences for risk reduction behaviors.
Impact of personalized risk information | 3 month
  Assess the impact of personalized risk communication to patients at risk for stroke on patient knowledge, beliefs, and preferences for risk reduction behaviors.

SECONDARY OUTCOMES:
Evaluate impact on medication adherence | 3-months
  Evaluate the impact of personalized risk communication on medication adherence at 3-months

CONTACTS AND LOCATIONS:
Overall Officials: Hayden Bosworth, PhD, Principal Investigator — Durham VA Medical Center
Locations (1):
- Durham VA Medical Center, Durham, North Carolina, United States

REFERENCES:
- [Derived] Powers BJ, Danus S, Grubber JM, Olsen MK, Oddone EZ, Bosworth HB. The effectiveness of personalized coronary heart disease and stroke risk communication. Am Heart J. 2011 Apr;161(4):673-80. doi: 10.1016/j.ahj.2010.12.021. PMID 21473965